CLINICAL TRIAL: NCT03667495
Title: Postoperative Oral and Intestinal Flora Changes in Patients With Colorectal Cancer and the Relationship Between These Changes and Prognosis
Brief Title: The Relationship Between Postoperative Changes of Oral and Intestinal Flora and Prognosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Yunwei Wei 2018-09-04
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Gut Microbiota; Oral Microbiota; Colorectal Cancer
Keywords: microbiota; colorectal cancer; recurrence
MeSH Terms: conditions — Colorectal Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Human fecal, oral and mucosal samples for DNA extraction.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Relapse: Patients who suffered colorectal cancer or adenoma relapse after curative surgery
- Remission: Patients who get remission after curative surgery

SUMMARY:
Specific oral microbiome has been found to contribute to the development of colorectal cancer. We speculate that specific oral microbiota related to colorectal cancer relapse after curative treatment. This study aim to discover if any difference of oral microbiota exist in patients who suffer from cancer relapse compared with patients who do not. Finally develop patient-centred programmes of surveillance protocols base on microbiota analysis.

DETAILED DESCRIPTION:
Colorectal cancer is a major cause of cancerrelated deaths and the third most commonly diagnosed cancer worldwide.Current estimates indicate that 20-30% of those who undergo treatment will experience recurrence and 35% of all patients will die within 5 years.

The human colon plays host to a diverse and metabolically complex community of microorganisms. While the specific oral microbiome has been found to contribute to the development of colorectal cancer. Investigators speculate that specific oral microbiota related to colorectal cancer relapse after curative treatment.

Patients are routinely offered surveillance in order to detect disease recurrence at an early, asymptomatic stage, with the intention of improving survival. Nevertheless, controversy continues to surround the optimal surveillance protocols. Investigators aim to discover if any difference of oral microbiota is exist in patients who suffer from relapse compared with patients who do not.

Future surveillance after colorectal cancer treatment should focus on risk-stratification. Finally investigators will develop patient-centred programmes of surveillance protocols base on microbiota analysis.

ELIGIBILITY:
Inclusion Criteria:

* Requirements of informed consent and assent of participant, parent or legal guardian as applicable
* Patients who underwent exhaustive colorectal cancer surgical resection and accept colonoscopy
* Patients between the age of 35 and 75 years old without considering sex
* Patients with BMI= 18.5-23.9
* Participants can follow the visit plan

Exclusion Criteria:

* Patients with colorectal cancer with distant metastasis
* Chronic renal diseases and hepatic cirrhosis
* Chronic ischemic heart disease with unstable angina, chronic heart failure at class III or IV and acute myocardial infarction in the last 6 months
* Individuals with a history of Chronic diarrhea
* Individuals with a history of Diabetes mellitus
* Individuals with a history of Hypertension
* Individuals with a history of autoimmune diseases
* Use of antibiotics and probiotics 3 mouth before samples collection
* Individuals with a history of abdominal operation due to any reason
* Individuals with any history of cancer other than colorectal cancer
* Individuals with Inflammatory bowel disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants were included according to the inclusion and exclusion criteria. Participants underwent an exhaustive colorectal cancer surgical resection in the First Affiliated Hospital of Harbin Medical University from September 1, 2017 to April 1, 2019. Participants did not use antibiotics and probiotics 3 mouth before samples collection.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-11-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Colorectal cancer or adenoma recurred | 12 months after surgery
  Use colonoscopy to check for recurrence of colorectal cancer

CONTACTS AND LOCATIONS:
Overall Officials: Yunwei Wei, Study Director — First Affiliated Hospital of Harbin Medical University
Locations (1):
- Yunwei Wei, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No